CLINICAL TRIAL: NCT07079800
Title: A Temporal Variability Study of Remimazolam for General Anesthesia Induction and Maintenance
Status: Active, not recruiting | Type: Observational
Sponsor: Jie Chen (Other)
Responsible Party: Sponsor-Investigator, Jie Chen, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Organization: The Second Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2025-120
Record Dates: First submitted 2025-06-18; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Biological Rhythm; Drug Metabolism and Pharmacokinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Remimazolam blood concentration and dosage measurement experiment Morning group
- Remimazolam blood concentration and dosage measurement experiment Afternoon group
- Remimazolam metabolic enzyme CES1 activity measurement experiment morning group
- Remimazolam metabolizing enzyme CES1 activity measurement experiment afternoon group

SUMMARY:
The purpose of this study was to observe and compare the differences in plasma concentration, dosage and carboxylesterase 1 activity of remimazolam when remimazolam is used for general anesthesia induction and maintenance at different times of the day, and to explore the effect of time rhythm on the pharmacokinetics and pharmacodynamics of remimazolam, so as to provide new ideas and clinical basis for optimizing medication regimens and anesthesia management.

DETAILED DESCRIPTION:
This study is a single-blind, prospective cohort study. It is mainly divided into two parts: 1. Detection of the blood concentration and dosage differences of remimazolam: Patients who were scheduled to undergo laparoscopic cholecystectomy under general anesthesia were included. The patients were divided into the morning group (operation time 8:00-12:00) and the afternoon group (operation time 14:00-18:00) according to the operation time. The blood concentration of remimazolam after anesthesia induction was measured, and the influence of time rhythm on the pharmacokinetics of remimazolam was statistically analyzed. The dosage of remimazolam used during anesthesia maintenance was measured, and statistical analysis was conducted on whether there were dosage differences and the temporal rhythm of drug efficacy of remimazolam during the maintenance process. 2. CES1 Activity detection: Patients who were scheduled to undergo laparoscopic partial hepatectomy under general anesthesia were included. The research subjects were divided into the morning group (8:00-12:00) and the afternoon group (14:00-18:00) based on the liver tissue sampling time. The activity of carboxylate esterase 1 (CES1) in the normal tissues adjacent to liver cancer in patients at different time points was measured. Analyze the influence of time rhythm on the drug metabolism of remimazolam. The effects of time rhythm on the pharmacokinetics and pharmacodynamics of remimazolam were jointly verified from three aspects: blood drug concentration, drug dosage, and CES1 activity.

ELIGIBILITY:
Inclusion Criteria:

Experiment 1: Measurement Experiment of Remimazolam Blood Concentration and Dosage

1. Age 18-65 years old, ASAI-II class, BMI18.5-25kg/m^2;
2. Inpatients undergoing laparoscopic cholecystectomy;
3. The estimated time of operation is 1.5~2.5 hours;
4. Voluntary participation and signed informed consent.

Experiment 2: Remimazolam metabolic enzyme CES1 activity measurement experiment

1. Age 18-75 years old, ASAI-III class;
2. Inpatients undergoing laparoscopic partial hepatic resection;
3. Voluntary participation and signed informed consent.

Exclusion Criteria:

Experiment 1:Measurement Experiment of Remimazolam Blood Concentration and Dosage

1. Pregnant or lactating women;
2. Patients who are allergic to remazolam or contraindicated;
3. Patients who are dependent on or tolerant to opioids or have long-term alcoholism;
4. Serious cardiovascular system, respiratory system, liver and kidney diseases;
5. History of obstructive sleep apnea;
6. Mental disorders or neurological diseases;
7. Patients who participated in clinical trials of other drugs within the last 3 months;
8. The attending physician or researcher considers that there are other circumstances that are not suitable for participation in this study;
9. Refuse to participate in the study

Experiment 2: Remimazolam metabolic enzyme CES1 activity measurement experiment

1. Pregnant or lactating women;
2. Patients who are allergic to remazolam or contraindicated;
3. Patients who are dependent on or tolerant to opioids or have long-term alcoholism;
4. Serious cardiovascular system, respiratory system;
5. History of obstructive sleep apnea;
6. Mental disorders or neurological diseases;
7. Patients who participated in clinical trials of other drugs within the last 3 months;
8. The attending physician or researcher considers that there are other circumstances that are not suitable for participation in this study;
9. Refuse to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experiment 1: Measurement Experiment of Remimazolam Blood Concentration and Dosage
  1. Age 18-65 years old, ASAI-II class, BMI18.5-25kg/m^2;
  2. Inpatients undergoing laparoscopic cholecystectomy;
  3. The estimated time of operation is 1.5~2.5 hours;
  4. Voluntary participation and signed informed consent.
  Experiment 2: Remimazolam metabolic enzyme CES1 activity measurement experiment
  1. Age 18-75 years old, ASAI-III class;
  2. Inpatients undergoing laparoscopic partial hepatic resection;
  3. Voluntary participation and signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Remimazolam dosage | During the operation
  During the maintenance of anesthesia, adjust the infusion rate of remimazolam to maintain the BIS value at 40-60, and record the dosage of remimazolam
Remimazolam blood concentration | Within two weeks after the operation
  Arterial blood of 2 ml was collected immediately after the end of remimazolam infusion during the anesthesia induction period and 6 minutes after the end of infusion, respectively. After each sample collection, rinse the ductus arteriosus with 1 ml of normal saline. The blood sample was drawn into a plastic tube containing ethylenediaminetetraacetic acid and stored at 4℃. Centrifuge the blood sample within 10 minutes after collection. Transfer the supernatant plasma into a polypropylene tube within 15 minutes after separation and store it immediately at -20℃. Blood samples should be stored at -80℃ within 4 hours after collection. The blood concentration of remimazolam and the concentration of its metabolite CNS7054 were determined by ultra-performance liquid chromatography-tandem mass spectrometry within two weeks after blood collection.
CES1 activity | Within two weeks after the operation
  When a surgeon removes a liver tumor, 50 mg of normal liver tissue adjacent to the tumor is quickly taken. The liver tissue is rinsed with normal saline, dried with filter paper, and placed in a cryotube. It is then rapidly frozen in liquid nitrogen and stored in a -80 ° C refrigerator for subsequent determination of CES1 enzyme activity by enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No